CLINICAL TRIAL: NCT04901975
Title: Acute Imposition of Fontan Physiology in The Single Ventricle Patient: Effects on Fibrosis, Function and Drug Intervention
Brief Title: Fibrosis and the Fontan
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-017716; 1R01HL149139-01A1 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-05-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Single-ventricle
MeSH Terms: conditions — Univentricular Heart | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Spironolactone (Experimental): Children will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers immediately prior to the Fontan operation.
  All SV children will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers ~1 year after the Fontan operation.
  Spironolactone is a mild diuretic. Drug dosage will be those used clinically and per the CHOP formulary: 3 mg/kg/day in divided doses every 6-24 hours; the drug will be weight adjusted every ~0.5 kg with a maximum dosage of 200 mg/24 hours. Maximum single dose is 100 mg.
  Spironolactone administration will begin after the Fontan procedure in the hospital prior to discharge or at the first outpatient visit ~ 2 weeks after discharge.
  Interventions: Drug: Spironolactone
- Observational (No Intervention): Children will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers immediately prior to the Fontan operation.
  All SV children, whether they received spironolactone or not, will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers ~1 year after the Fontan operation. Demographics and medical history will be collected again along with adverse events. Children will also undergo CMR for evaluation of hemodynamics, ventricular function (including strain), computational modeling and lymphatic abnormalities. A few of these patients will be undergoing CMR for clinical reasons and study CMR related and study MRI related imaging and blood draws will be performed in coordination with their clinical care (ie these sequences will be added on to their clinical sequences).
- Control (No Intervention): The purpose of this study is to non-invasively characterize the fibrotic consequences of SV physiology, its possible solution and effect on lymphatics. This project investigates the response to acute imposition of Fontan hemodynamics by examining the interrelationship between liver and cardiac fibrosis/dysfunction and lymphatic congestion (figure 1) along with a pilot trial of the antifibrotic agent, spironolactone, to prevent these consequences and to determine if MRI can discern these differences. The combination of serum biomarkers and MRI form a powerful non-invasive tool in putting together this complicated web of dysfunction.
  Control subjects who are non-SV patients but who have normal heart function who are undergoing CMR for evaluation (eg patients undergoing CMR for vascular ring evaluation, family history of congenital heart disease but found to be normal, etc) will have study related MRI and CMR sequences performed.
- Observational - 1A (No Intervention): Subjects who were enrolled in this study in Spironolactone arm and patient's family would like to continue participation.
  All SV children, whether they received spironolactone or not, will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers ~1 year after the Fontan operation. Demographics and medical history will be collected again along with adverse events. Children will also undergo CMR for evaluation of hemodynamics, ventricular function (including strain), computational modeling and lymphatic abnormalities. A few of these patients will be undergoing CMR for clinical reasons and study CMR related and study MRI related imaging and blood draws will be performed in coordination with their clinical care (ie these sequences will be added on to their clinical sequences).
- Observational - 1B (No Intervention): Subjects who were enrolled in other studies with intervention.
  All SV children, whether they received spironolactone or not, will undergo characterization and measurement of liver and cardiac fibrosis with MRI and cardiac magnetic resonance (CMR) as well as serum biomarkers ~1 year after the Fontan operation. Demographics and medical history will be collected again along with adverse events. Children will also undergo CMR for evaluation of hemodynamics, ventricular function (including strain), computational modeling and lymphatic abnormalities. A few of these patients will be undergoing CMR for clinical reasons and study CMR related and study MRI related imaging and blood draws will be performed in coordination with their clinical care (ie these sequences will be added on to their clinical sequences).

INTERVENTIONS:
Drug: Spironolactone — Spironolactone is a mild diuretic. Drug dosage will be those used clinically and per the CHOP formulary: 3 mg/kg/day in divided doses every 6-24 hours; the drug will be weight adjusted every ~0.5 kg with a maximum dosage of 200 mg/24 hours. Maximum single dose is 100 mg. Spironolactone, the aldosterone antagonist to be utilized in Specific Aim 2 of this study, is FDA approved, has been on the market for many years and is routinely administered to all types of children with congenital heart disease including SV patients. The choice of which patient this should be administered to is up to the clinician and their patients and therefore, not all SV patients are on this medication.
  Arms: Spironolactone

SUMMARY:
The purpose of this study is to non-invasively characterize the fibrotic consequences of single ventricle physiology, its possible solution and effect on lymphatics. This project investigates the response to acute imposition of Fontan hemodynamics by examining the interrelationship between liver and cardiac fibrosis/dysfunction and lymphatic congestion along with a pilot trial of the antifibrotic agent, spironolactone, to prevent these consequences and to determine if MRI can discern these differences. The combination of serum biomarkers and MRI form a powerful non-invasive tool in putting together this complicated web of dysfunction.

DETAILED DESCRIPTION:
Fontan patients, unfortunately, suffer multiple complications such as liver fibrosis, cardiac fibrosis and lymphatic congestion. While investigations describing the clinical state are taking place in older children and young adults, the onset of these complications remains unclear. The knowledge gap this proposal seeks to fill is understanding how early liver and cardiac fibrosis develops as well as lymphatic abnormalities by assessing these before as well as early after imposition of the Fontan circulation.

Single ventricle case subjects will be between aged 1 and less than or equal to 6 years of age of either gender, whether single left or right ventricle, who are scheduled to undergo a Fontan operation at the Children's Hospital of Philadelphia (CHOP) and control subjects will be aged between 1 and less than or equal to 6 years of age with normal ventricular function and normal livers who present to CHOP for a clinically indicated MRI.

Review of medical records, demographic/social history, physical examination (performed for clinical purposes), administer study drug (spironolactone), blood tests (serum biomarkers), MRI/CMR (including a non-FDA approved MRI sequence), liver assessment, administration of contrast and general anesthesia for case subjects (in some instances, an extension of clinically indicated anesthesia for control and some case subjects approximately 15-20 minutes) as applicable.

The difference between enrollment and 1 year after Fontan surgery for a) liver fibrosis measured by Magnetic Resonance Elastography (MRE) and T1 mapping, b) cardiac fibrosis measured by T1 mapping using global extracellular volume (ECV) and c) percentage of myocardial mass which demonstrates delayed enhancement (DE). This is for both non-drug and spironolactone administered groups

ELIGIBILITY:
Inclusion Criteria:

* Single Ventricle (SV) Patients

Cohort 1 (Observational Group - no study medication):

* Subjects between 1 and ≤ 6 years of age of either gender.
* Either single left or single right ventricle.
* Subjects who are scheduled to undergo a Fontan operation at CHOP.
* Parents signing informed consent.

Cohort 1A (formerly part of study drug group who wish continued participation in the observational group):

* Subjects who were enrolled in this study in Cohort 2 and are either non-compliant with the medication, no longer want to take the medication, or have an AE that requires them to stop the medication, and patient's family would like to continue participation
* Patients were on study medication for 6 weeks or less.
* The principal investigator deems it appropriate for the patient to switch to the observational arm.
* Patients signing the observational informed consent form.

Cohort 1B (observational group - in other studies with intervention):

* Subjects between 1 and ≤6 years of age of either gender.
* Either single left or single right ventricle.
* Subjects who are planned to undergo a Fontan operation at CHOP.
* Patients in other interventional studies approved by principal investigator.
* Patients signing the observational informed consent form.

Cohort 2 (study drug Group - spironolactone):

* Subjects between 1 and ≤ 6 years of age of either gender.
* Either single left or single right ventricle.
* Subjects who are scheduled to undergo a Fontan operation at CHOP.
* Parents signing informed consent.

Controls

* Subjects between 1 and ≤ 6 years of age of either gender
* Subjects with normal ventricular function and normal livers who present to CMR for clinical indications and require anesthesia.
* Receiving contrast for clinical purposes. No control patient will receive contrast for research purposes.
* Parents signing informed consent.

Exclusion Criteria:

-

Cohort 1 (Observational Group - no study medication):

* Subjects with any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contradiction to a sedated CMR (i.e. presence of a pacemaker).
* Patient currently taking spironolactone or eplerenone
* Subjects in any study that would preclude participation in the study by altering results

Cohort 1A (formerly part of study drug group who wish continued participation in the observational group):

* Subjects with any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contradiction to a sedated CMR (i.e. presence of a pacemaker).
* Subjects in any study that would preclude participation in the current study.

Cohort 1B (observational group - in other studies with intervention):

* Subjects with any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contradiction to a sedated CMR (i.e. presence of a pacemaker).
* Patient currently taking spironolactone or eplerenone
* Subjects in any study that would preclude participation in the current study or studies not approved by principal investigator.

Cohort 2 (Study Drug Group - Spironolactone):

* Subjects with any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contradiction to a sedated CMR (i.e. presence of a pacemaker).
* Patient currently taking spironolactone or eplerenone
* Subjects with hyperkalemia or Addison disease;
* Subjects on enalapril or other angiotensin receptor blockers
* Subjects with a history of hypersensitivity to spironolactone suspension or any component of the formulation
* Subjects with a clinically documented diagnosis of severe renal insufficiency (implying estimated glomerular filtration rate (eGFR) <30 mL/minute/1.73 m2).
* Subjects in any study that would preclude participation in the study by altering results

Controls

* Any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
* Any contradiction to a sedated CMR (i.e. presence of a pacemaker).
* Patient currently taking spironolactone, eplerenone or an angiotensin converting the enzyme inhibitor/angiotensin receptor blocker.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Liver elastography by MRE prior to and after Fontan | up to 1 year
  Measured by MRE for viscoelastic properties of the liver, primarily stiffness
Liver elastography by T1rho prior to and after Fontan | up to 1 year
  Measured by T1rho mapping for further viscoelastic properties of the liver, primarily hepatic fibrosis
Heart tissue characterization by T1 mapping prior to and after Fontan | up to 1 year
  Measured by T1 mapping using global extracellular volume (ECV)
Heart tissue characterization prior to and after Fontan | up to 1 year
  Percentage of myocardial mass which demonstrates delayed enhancement

SECONDARY OUTCOMES:
Serum biomarkers of fibrosis | up to 1 year
  Serum biomarkers of liver will be assessed to include eg Galectin-3, PIIIP and TGF-beta
Lymphatic dysfunction by MRE prior to and after Fontan | up to 1 year
  Lymphatic dysfunction will be measured by MRE to find if lesions are present
Lymphatic dysfunction T1rho prior to and after Fontan | up to 1 year
  Lymphatic dysfunction will be measured by T1rho to find if lesions are present

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fogel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No